CLINICAL TRIAL: NCT04586829
Title: The Effect of Two Dietary Interventions on the Symptomatic Control of People Living With Anxiety Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Luis Adrian Soto Mota, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UIE-3506-20-21-1
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional diet (Active Comparator): Conventional diet. (50% carbohydrate, 30% lipids, 20% protein). Current dietary recommendations from official guidelines will be reinforced.
  Interventions: Other: Diet
- Ketogenic diet (Experimental): Tailored ketogenic diet. Participants will be allowed to chose their meals as long as they consume less than 50gr of carbohydrates per day.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — <50 grams of total carbohydrates per day. Monosaturated fats consumption will be encouraged over saturated fats.

SUMMARY:
This randomised controlled trial will evaluate the effect of a ketogenic diet vs a conventional diet on the symptoms of patients living with anxiety disorders using a validate self-reported inventory.

DETAILED DESCRIPTION:
It has been theorized that ketogenic diet could improve symptom control in patients living with anxiety disorders. Animal models support this hypothesis but to this date, studies in humans are lacking.

The investigators will randomise patients with a confirmed diagnosis of anxiety disorders to follow a ketogenic diet (<50 grs of carbohydrate per day) or a conventional diet (50% carbohydrate, 30% lipids, 20% protein) for one month.

Symptom control will be assessed weekly using Beck's inventory for Anxiety. Diet adherence will be measured using standardised food frequency logs and acetoacetate urine strips.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Anxiety Disorder by Psychiatrist.

Exclusion Criteria:

* Patients with the diagnosis of drug abuse, cognitive impairment or dementia, porphyria, carnitine translocase deficiency and carnitine palmitoyl transferase deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Symptom control | One month
  Total points in Beck's Inventory for Anxiety. Scores range between 0 to 63 and higher numbers mean a worse outcome.

SECONDARY OUTCOMES:
Subjective self perceived control | One month
  Self-assessed and reported symptom ranging between 0 - 100. Higher numbers mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Soto, MD,DPhil, Principal Investigator — Biomedical Sciences Researcher
Locations (1):
- INCMNSZ, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Upon request to PI.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after publication
Access Criteria: Send email to adrian.sotom@incmnsz.mx

REFERENCES:
- [Background] Ari C, Kovacs Z, Juhasz G, Murdun C, Goldhagen CR, Koutnik AP, Poff AM, Kesl SL, D'Agostino DP. Corrigendum: Exogenous Ketone Supplements Reduce Anxiety-Related Behavior in Sprague-Dawley and Wistar Albino Glaxo/Rijswijk Rats. Front Mol Neurosci. 2017 Feb 13;10:36. doi: 10.3389/fnmol.2017.00036. eCollection 2017. PMID 28210213
- [Background] Fydrich, T., Dowdall, D. and Chambless, D. L. (1992) 'Reliability and validity of the beck anxiety inventory', Journal of Anxiety Disorders, 6(1), pp. 55-61. doi: 10.1016/0887-6185(92)90026-4.
- [Background] Kashiwaya Y, Bergman C, Lee JH, Wan R, King MT, Mughal MR, Okun E, Clarke K, Mattson MP, Veech RL. A ketone ester diet exhibits anxiolytic and cognition-sparing properties, and lessens amyloid and tau pathologies in a mouse model of Alzheimer's disease. Neurobiol Aging. 2013 Jun;34(6):1530-9. doi: 10.1016/j.neurobiolaging.2012.11.023. Epub 2012 Dec 29. PMID 23276384
- [Background] Kovacs Z, D'Agostino DP, Diamond D, Kindy MS, Rogers C, Ari C. Therapeutic Potential of Exogenous Ketone Supplement Induced Ketosis in the Treatment of Psychiatric Disorders: Review of Current Literature. Front Psychiatry. 2019 May 23;10:363. doi: 10.3389/fpsyt.2019.00363. eCollection 2019. PMID 31178772
- [Background] Saslow LR, Daubenmier JJ, Moskowitz JT, Kim S, Murphy EJ, Phinney SD, Ploutz-Snyder R, Goldman V, Cox RM, Mason AE, Moran P, Hecht FM. Twelve-month outcomes of a randomized trial of a moderate-carbohydrate versus very low-carbohydrate diet in overweight adults with type 2 diabetes mellitus or prediabetes. Nutr Diabetes. 2017 Dec 21;7(12):304. doi: 10.1038/s41387-017-0006-9. PMID 29269731
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538